CLINICAL TRIAL: NCT02499848
Title: Phase IIa Study, Evaluating the Safety and Tolerability of Targeted Intraprostatic Administration of PRX302 With Histologically Proven,Clinically Significant Localised, Low to Intermediate Risk Prostate Cancer Associated With MRI Lesion
Brief Title: Evaluate, Safety and Tolerability of Intraprostatic PRX302 Administration, Low to Intermediate Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sophiris Bio Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRX302-2-07
Record Dates: First submitted 2015-06-30; First posted 2015-07-16 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: MRI Lesion; transperineal injection; prostate biopsies
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PRX302

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraprostatic administration (Experimental): PRX302
  Interventions: Drug: PRX302

INTERVENTIONS:
Drug: PRX302 — Single prostate cancer lesion injected with PRX302.
  Other Names: Topsalysin

SUMMARY:
To Evaluate Safety, Tolerability and Potential Efficacy of PRX302 effect on clinically significant localised low to intermediate prostate cancer.

DETAILED DESCRIPTION:
A single center, open label, Phase IIa, Idea, Development, Exploration, Assessment, Long-term follow-up (IDEAL) prospective development study. The study will treat approximately 20 men who meet the eligibility criteria, and give written informed consent. Safety and Tolerability will be assessed post-treatment at 2 days (phone call), 2 weeks, 6 weeks, 12 weeks, 24 weeks and 26 weeks. Potential Efficacy will be assessed by biopsy at 24 weeks and imaging (MRI) at 2 weeks, 12 weeks and 24 weeks and PSA outcomes at 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥40 years and life expectancy of ≥10 years.
* Serum prostate-specific antigen (PSA) ≤15 ng/mL.
* Transperineal prostate biopsy within 12 months prior to dosing, with a clinically significant lesion correlating with an mpMRI visible lesion.
* Radiological stage T1-T2 N0 Mx/M0 disease.
* A visible lesion on mpMRI that is accessible to PRX302 transperineal injection.

Exclusion Criteria:

* Previous radiation therapy to the pelvis.
* Androgen suppression or anti-androgen therapy within the 12 months prior to dosing, for prostate cancer.
* Use of a 5-alpha reductase inhibitor within the 3 months prior to dosing.
* Evidence of metastatic disease or nodal disease outside the prostate on bone scan or cross-sectional imaging.
* Inability to tolerate a transrectal ultrasound (TRUS).
* Known allergy to latex or gadolinium (Gd).
* Previous electroporation, radiofrequency ablation, high-intensity focused ultrasound (HIFU), cryosurgery, thermal or microwave therapy to treat cancer of the prostate.
* Unable to have pelvic MRI scanning (severe claustrophobia, permanent cardiac pacemaker, metallic implant, etc. likely to contribute significant artifact to images).

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of a single injection of PRX302 in all patients will be assessed by recording Adverse Event assessments over 24 weeks | Week 24

SECONDARY OUTCOMES:
To evaluate the potential efficacy of PRX302 by • Transperineal targeted biopsy performed of the treated area at 24 weeks post-treatment | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Hashim U Ahmed, PhD,FRCS, Principal Investigator — Division of Surgery & Interventional Science University College London
Locations (1):
- UCLH, London, United Kingdom